CLINICAL TRIAL: NCT05536648
Title: "Comparing the Plaque Removal Ability of Triple Head Tooth Brush Versus Single Head Tooth Brush Among School Based Cerebral Palsy Children:A Randomized Control Trial"
Brief Title: "Comparing the Plaque Removal Ability of Two Different Toothbrushes Among School Going CP Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Zainab Jahanzeb, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DowUHS clnical trial
Record Dates: First submitted 2022-09-05; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Cerebral Palsy
Keywords: plaque status; difficulties assocaited with tooth brushing; triple head tooth brush
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: single blinded randomized control trial
Who Masked: Investigator
Masking Description: The dental investigator who perform the oral health assessment for dentition status and plaque status was blinded during the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Single head toothbrush (Experimental): Cerebral palsy children were given single head tooth brush along with fluoridated toothpaste for brushing.
  Interventions: Other: Comparing the plaque removal ability of triple head tooth brush versus single head tooth brush among school based cerebral palsy children: A Randomized Control Trial
- Group 2 Triple head toothbrush (Experimental): Cerebral palsy children were given triple head tooth brush along with fluoridated toothpaste for brushing.
  Interventions: Other: Comparing the plaque removal ability of triple head tooth brush versus single head tooth brush among school based cerebral palsy children: A Randomized Control Trial

INTERVENTIONS:
Other: Comparing the plaque removal ability of triple head tooth brush versus single head tooth brush among school based cerebral palsy children: A Randomized Control Trial — To compare the plaque removing ability of two different tooth brushes in school going cerebral palsy children.

SUMMARY:
It was an intervention utilizing two toothbrushes on school going cerebral palsy children age (6 -18 yrs). The triple head tooth brush and single head brush was provided to parents along with dental health education to their parent on brushing technique and oral care for their child. Parents who give consent for their child were enrolled in the study. The plaque removal ability of toothbrush was assessed by Turesky modified Quigley Hein index. The reading for plaque score was recorded at base line and after the follow up of 4 weeks. Difficulties during brushing was also analyzed.

DETAILED DESCRIPTION:
Study Design :Single blinded Randomized Control Trial

Study Setting: The study was conducted in schools that have cerebral palsy children in Karachi.

Study Duration :From June 2021 to June 2022.

Sampling technique: Non probability purposive sampling technique was used for selection of study population.

Sample Size: Total 58 individuals were recruited in the study. After including the 20% drop out rate 35 subjects were enrolled at each study group which make total sample size of 70 Cerebral Palsy participants. Random allocation was made in two groups in order to keep the sizes of intervention groups similar.

Study Instrument:

* For study intervention two types of tooth brushes were used. The single head and triple head tooth brush.
* For data collection a structured questionnaire was used that collect information on social demographic characteristics, oral hygiene behavior, dentition status, plaque status and difficulties associated with brushing.

Data Collection Method:

* The study used a single-blind, parallel, and randomized controlled trial (RCT) design.
* A total 70 Cerebral palsy children were recruited in the study which was stratified into two groups of 35 children each in intervention and control group.
* Intervention group was given triple head tooth brush with fluoridated toothpaste whereas control group was given single head tooth brush with fluoridated toothpaste.
* Dental health education on oral care was given to participant's parent along with brushing technique demonstrated on model as well on their child's teeth.
* Data was collected through structured questionnaire. Oral health assessment was recorded through DMFT/dmft index. Plaque index was calculated by Turesky modified Quigley Hein index by dyeing the plaque on tooth surface by plaque disclosing tablets. Difficulties during brushing were also evaluated.
* Statistical analysis involved pair sample t test, repeated measure ANOVA, Chi-square and Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* • Parents who give consent to enrol in study and their children (age: 6-18yrs) who cooperate to allow to perform oral assessment.

Exclusion Criteria:

* • Children unable to cooperate due to underlying systematic condition because of their motor and mental illness.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Plaque Index Score | Before and after the intervention of four weeks
  Plaque score was recorded through Turesky modified Quigley Hein Index to observe improvement in plaque score before and after the intervention.
Difficulties associated with toothbrushing e.g Bleeding during brushing, gag reflex, enable reaching more teeth and time required for brushing. | At postintervention after four weeks.

SECONDARY OUTCOMES:
DMFT/dmft index | At Baseline
  To assess dentition status
Oral Hygiene Behavior e.g. brushing frequency, complain of pain and visit to a dentist during last 12 months | At Baseline
  Brushing frequency, complain of pain and visit to a dentist during last 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Shah, M.Sc,Mphil, Study Chair — Dow University of Health Sciences
Locations (1):
- Zainab Khaliq Ansari, Karachi, Sindh, Pakistan